CLINICAL TRIAL: NCT01141959
Title: Blood Samples to Identify Biomarkers in Haploidentical Graft Recipients
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: FHCRC-2373.00; IR-7093 (Other: FHCRC); R01HL091744-02S1 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-11 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2015-03

CONDITIONS: Leukemia; Hodgkin Disease; Non-Hodgkin Lymphoma; Myelodysplastic Syndrome; Multiple Myeloma
Keywords: hematopoietic stem cell transplantation; cyclophosphamide; fludarabine; mycophenolate mofetil; mycophenolic acid; biomarkers
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are interested in identifying patient-specific factors related to donor chimerism in patients who receive nonmyeloablative hematopoietic stem cell transplants from haploidentical donors. We will look how patients' bodies break down and immediately respond to cyclophosphamide, fludarabine and mycophenolate mofetil.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive nonmyeloablative conditioning which includes fludarabine
* Scheduled to receive a haploidentical graft
* Scheduled to receive postgrafting immunosuppression which includes oral mycophenolate mofetil (MMF) or enteric-coated mycophenolic acid
* Age >18 years at the time of enrollment

Exclusion Criteria:

* Diagnosed with an immunodeficiency disorder, including HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematopoeitic cell transplant patients with haploidentical donors receiving cyclophosphamide, fludarabine and mycophenolate mofetil.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Donor T-cell chimerism | Day 28 post-transplant

SECONDARY OUTCOMES:
Exposure to cyclophosphamide, fludarabine, and mycophenolate mofetil and their breakdown products | 1 week before through 3 weeks after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine McCune, PharmD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States